CLINICAL TRIAL: NCT05321667
Title: Patients Without Standard Modifiable Cardiovascular Risk Factors (SMuRF-less) and Their Prognosis After a ST-segment-Elevation Myocardial Infarction (STEMI)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Batric POPOVIC, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2021PI154
Record Dates: First submitted 2022-03-26; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: STEMI
Keywords: SMuRFs; SMuRF-less; Standard Modifiable Risk Factors; Prognosis; Family History
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMuRF-less: Patients presenting no standard modifiable risk factor of cardiovascular disease (diabetes mellitus, hyperlipidemia, hypertension, and cigarette smoking).
- SMuRFs: Patients presenting at least one standard modifiable risk factor of cardiovascular disease (diabetes mellitus, hyperlipidemia, hypertension, and cigarette smoking).

SUMMARY:
The purpose of this study is to asses the prognosis of STEMI patients without standard modifiable risk factors of cardiovascular disease (diabetes mellitus, hyperlipidemia, hypertension and cigarette smoking) compare to patients presenting at least one of these risk factors.

ELIGIBILITY:
Inclusion Criteria:

STEMI patients who had a percutaneous coronary intervention (PCI) in our PCI center.

Exclusion Criteria:

Pain duration exceeding 24h. Perioperative STEMI, including STEMI related to cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systematic review of STEMI patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
MACE (Major Adverse Cardiovascular Event) | 3 years
  Composite outcome including cardiovascular death or incidence of acute coronary syndrome, ischemic stroke or heart failure.

SECONDARY OUTCOMES:
All-cause mortality | 3 years
Number of patients presenting cardiovascular death during the follow-up | 3 years
  Number of patients presenting death due to fatal myocardial infarction, fatal ischemic stroke, sudden death, severe heart failure and cardiogenic shock during the follow-up.
Number of patients presenting heart failure during the follow-up | 3 years
  Number of patients hospitalized for acute heart failure during the follow-up, as well as patients presenting persistent symptoms of chronic heart failure after their STEMI (dyspnea NYHA > 1) and/or long-terme need for diuretics.
Number of patients presenting ischemic stroke during the follow-up | 3 years
  Number of patients presenting fatal or non fatal ischemic stroke during the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du Coeur et des Vaisseaux Louis Mathieu, Vandœuvre-lès-Nancy, Meurthe-et-Moselle, France